CLINICAL TRIAL: NCT06005974
Title: A Phase 2, Open Label Study of REC-4881 in Participants With Unresectable Locally Advanced or Metastatic Cancer With AXIN1 or APC Mutation
Brief Title: A Study of REC-4881 in Participants With Cancers Which Have an AXIN1 or APC Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to sponsor decision. This decision was not related to safety concerns.
Sponsor: Recursion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-4881-221
Record Dates: First submitted 2023-08-10; First posted 2023-08-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: AXIN1 Gene Mutation; APC Gene Mutation; Solid Tumor
Keywords: AXIN1; APC; Locally advanced or metastatic; Solid tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Participants are allocated to two groups, AXIN1 mutation or APC mutation, in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXIN1 Cohort (Experimental): Participants will receive REC-4881 12mg PO dosed QD
  Interventions: Drug: REC-4881
- APC Cohort (Experimental): Participants will receive REC-4881 12mg PO dosed QD
  Interventions: Drug: REC-4881

INTERVENTIONS:
Drug: REC-4881 — REC-4881 4mg capsules

SUMMARY:
This is a multi-center, open-label study to investigate the safety, efficacy and pharmacokinetics of REC-4881 (12 mg PO daily doses) for the treatment of participants with unresectable locally advanced or metastatic solid tumors with AXIN1 or APC mutation.

ELIGIBILITY:
Inclusion Criteria:

1. 55 years of age or older with histologically-confirmed unresectable, locally advanced, or metastatic solid tumor with AXIN1 or APC mutation. If a participant has colorectal cancer, then they must be RAS / RAF wild type to enroll into the APC mutant cohort
2. Have experienced progressive disease, relapsed disease, or be intolerant to at least one established standard systemic anti-cancer treatment, or in the opinion of the Investigator have been considered ineligible for standard therapy
3. Measurable disease at baseline per RECIST 1.1 criteria
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

1. Received treatment with another mitogen-activated protein kinase (MEK) inhibitor within two months of first dose of REC-4881
2. Left ventricular ejection fraction (LVEF) <50% as measured by echocardiogram (ECHO) or multigated acquisition (MUGA) scan

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities | Up to 24 months
Objective Response Rate | Up to 24 months

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of REC-4881 | pre-dose and up to 24 months
Disease Control Rate | Up to 24 months
Duration of response | Up to 24 months
Duration of Stable Disease | Up to 24 months
Time to Response | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Sharp Memorial Hospital, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Mission Cancer And Blood, Des Moines, Iowa
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Saint Luke's Hospital, Kansas City, Missouri
  - Hunterdon Hematology Oncology, Hillsborough, New Jersey
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No